CLINICAL TRIAL: NCT06674109
Title: SAVE-Care (SGLT2i As Novel Gout Care) Trial
Brief Title: SAVE-Care (Sodium Glucose Cotransporter-2 Inhibitors [SGLT2i] As Novel Gout Care) Trial
Acronym: SAVE-Care
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hyon Choi, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2024P003219; 1R61AR084188-01A1 (NIH)
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Gout and Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Empagliflozin 10mg (Experimental): Participants in this arm will take empagliflozin 10mg daily
  Interventions: Drug: Empagliflozin 10 mg
- Placebo (Placebo Comparator): Participants in this arm will take a placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 mg — For the empagliflozin arm, participants will take 10 mg daily.
  Other Names: Jardiance
  Arms: Empagliflozin 10mg
Drug: Placebo — Participants in the placebo arm will take a placebo daily.
  Arms: Placebo

SUMMARY:
SAVE-Care (Sodium Glucose Cotransporter-2 inhibitors [SGLT2i] As Novel Gout Care) Trial is a double-blind randomized placebo-controlled trial (RCT) designed to assess the effect of empagliflozin on serum urate [SU] levels of gout patients, as well as levels of highly-sensitivity C-reactive protein [hsCRP] and interleukin 6 [IL-6], and estimate gout flares over 3 months, in order to develop a full-scale RCT of clinical endpoints to directly inform gout care guidelines.

DETAILED DESCRIPTION:
With the compelling premise as above, prospective gout-patient-specific RCTs for key gout disease endpoints are needed to provide high-level evidence needed to impact practice change with a great likelihood to revolutionize gout care as SGLT2i did in cardiology, diabetology, and nephrology. To that end, the investigators propose to conduct the first RCT of SGLT2i specifically among gout patients with hyperuricemia (SAVE-Care [SGLT2i As Novel Gout Care] Trial) for the endpoint of serum urate, the central outcome in clinical care, trials, and FDA approvals, as discussed above. Specifically, the investigators will conduct a double-blind RCT of 60 gout patients, with 2 parallel arms of empagliflozin 10mg daily vs. placebo in a 2:1 ratio over 12 weeks.

The SAVE-Care trial will fill an important evidence gap by determining the magnitude of SU reduction specifically in patients with well-characterized gout, and with hyperuricemia and recent flares, for whom gout treatment would be indicated. If SU reduction is substantial (e.g. >~1.5mg/dL) as hypothesized in Aim 1, SGLT2i will be considered a useful urate-lowering gout therapy given their proven cardiovascular [CV]-kidney-metabolic benefits, particularly for typical cases managed by primary care or those with indicated CV-kidney metabolic comorbidities. However, if the urate-lowering capacity among gout patients is relatively small, SGLT2i's clinical utility for SU control purpose (vs flare control alone) will be considered limited. To that end, SU outcomes data generated by the SAVE-Care trial in relevant gout patients will be directly applicable to clinical gout care.

The SAVE-Care trial will also provide first prospective RCT outcomes data on two relevant inflammatory markers (i.e., hs-CRP and IL-6) among gout patients to assess the anti-inflammatory potentials of SGLT2i relevant to gout. Furthermore, SAVE-Care trial will generate estimates for gout flare risks and rates in the empagliflozin and in the placebo group over 12 weeks, which will serve as important preliminary data to developing a future full-scale RCT for clinical endpoints. All in all, with the overarching goal of improving gout outcomes and its comorbidities together, this study will not only generate immediately actionable evidence on the central outcome of SU, the causal biomarker of gout, but also key data on inflammatory markers, flares, and medication adherence in SGLT2i and placebo to inform future trials.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form.
2. Fulfilling American College of Rheumatology [ACR]/European Alliance of Associations for Rheumatology [EULAR] gout criteria
3. 1+ gout flares in last 12 months
4. Serum urate level ≥ 6mg/dl
5. Males and females; Age 18-80
6. Willingness to adhere to the study intervention procedures.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Estimated Glomerular Filtration Rate [eGFR] <20ml/min
2. Colchicine or nonsteroidal anti-inflammatory drug [NSAID] prophylaxis
3. active cardiovascular disease [CVD], type-1 diabetes
4. pregnant and lactating women
5. Presence of a condition(s) or diagnosis, either physical or psychological, or physical exam finding that precludes participation. [History of ketoacidosis, end-stage or decompensated liver disease, active cancer]
6. Use of anti-obesity drugs
7. Basal-bolus or multiple daily injection insulin regimens, or loop diuretics

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Serum Urate Change | Screening to three months of follow-up
  Change in serum urate [SU] levels as compared with controls at Week 12. SU levels will be obtained at screening and Week 4, 8, and 12.

SECONDARY OUTCOMES:
Changes in highly selective C-reactive protein (hsCRP) | Screening to three months of follow-up
  hs-CRP levels will be measured at screening and Week 12
Gout flares | Screening to three months of follow-up
  Gout flares will be ascertained using the Gaffo criteria, which requires presence of three or more out of the four items included in the flare diary and asked at each study visit: 1) subject-defined gout-flare, 2) pain at rest >3 on a 0-10 numeric scale, 3) presence of at least one swollen joint, and 4) presence of at least one warm joint.
Medication Adherence | Baseline to three months of follow-up
  Adherence to empagliflozin or placebo, defined by taking 80% or more of the dispensed doses and calculated by the number of pills taken (pills dispensed - pills counted).
Changes in Interleukin 6 [IL-6] | Screening to three months of follow-up
  IL-6 levels will be measured at screening and 12 weeks.

OTHER OUTCOMES:
Quality of Life Measures (36-Item Short Form Survey) | Screening to two months of follow-up
  The 36-Item Short Form Survey [SF-36] will be administered at screening and eight weeks later to measure quality of life measures
Quality of Life Assessment [GAQ] | Screening to three months after baseline
  The Gout Assessment Questionnaire [GAQ] will be administered at screening and every monthly visit for the full three month period to assess quality of life in specific regards to gout outcomes.
Tophi Measurement | Screening
  If tophi are present in participants at screening, tophi will be measured for the maximum diameter of the longest tophus using a Vernier caliper and the total number and sites of tophi.
Work Productivity and Activity Impairment Questionnaire [WPAI] | Screening to three months of follow-up
  Participant absences from work and other work-related outcomes will be measured at every visit from screening to the final visit twelve weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Hyon K Choi, MD, DrPH, Principal Investigator — Massachusetts General Hospital